CLINICAL TRIAL: NCT02345967
Title: Function of Implanted Glucose Sensor 2
Acronym: FIGS-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlySens Incorporated (Industry)
Collaborators: Profil Institute for Clinical Research, Inc. (Other); AMCR Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PR13-004
Record Dates: First submitted 2015-01-20; First posted 2015-01-26 (Estimated); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Diabetes Mellitus
Keywords: diabetes mellitus requiring insulin
MeSH Terms: conditions — Diabetes Mellitus

ARMS (1):
- Study Group (Experimental): Device: Model 100 Sensor
  Interventions: Device: Model 100 Sensor

INTERVENTIONS:
Device: Model 100 Sensor — One Model 100 Sensor to be implanted per subject.

SUMMARY:
The purpose of this study is to verify safety and assess tolerance of a long-term, implanted glucose monitoring sensor. The study will also provide data to characterize the response properties and calibration of the implanted sensor and determine if such properties vary with implant duration.

ELIGIBILITY:
Inclusion Criteria:

* Either: (1) male or (2) female and not pregnant, breastfeeding, or planning to become pregnant
* Diabetes diagnosis of type 1, or type 2 using insulin
* Under the routine care of a physician for diabetes treatment
* Able to understand and follow directions
* History of compliance with diabetes care regimen
* Able to comply with study requirements regarding planned clinical visits and exams
* In good physical condition without major medical concerns or blood chemistry abnormalities

Exclusion Criteria:

* Mental disorders that might affect compliance to protocols
* Diabetes diagnosis type 2 where treatment involves (1) oral medication without insulin or (2) insulin use restricted to a single daily injection of long-acting insulin or (3) control by diet/exercise regimen alone
* History of intolerance or sensitivity to any of the device materials
* History of any adverse reaction or allergy to any of the drugs/agents utilized in the study procedures
* History of recurrent skin infections

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01; Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | From enrollment to 2-weeks post-explant
  Incidence of adverse events related to the Intervention

CONTACTS AND LOCATIONS:
Overall Officials: Linda Morrow, MD, Principal Investigator — Profil Institute for Clinical Research, Inc.
Locations (2):
- United States (2):
  - Profil Institute for Clinical Research, Chula Vista, California
  - AMCR Institute, Escondido, California